CLINICAL TRIAL: NCT04148027
Title: Use of Telemedicine for Geriatric Emergency Patients
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Dr. Oliver Matz, Consultant, RWTH Aachen University
Other Study IDs: Telenotfallgeriatrie-2017; EK 243/17 (Other: local ethics committee)
Record Dates: First submitted 2019-10-28; First posted 2019-11-01 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Geriatric Patients
Keywords: emergency medicine; geriatrics; telemedicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Treatment recommendation by emergency department physicians — Standard treatment after admission in the emergency department from a team of residents in internal medicine, neurology and general surgery.
Other: Treatment recommendation by telemedical geriatric co-evaluation — Treatment recommendation from a board-certified geriatrician linked for co-evaluation by means of video transmission

SUMMARY:
The aim of the present study is the implementation of a telemedical geriatric co-evaluation in the area of the emergency department. The use of telemedicine is intended to improve the care of geriatric emergency patients.

Primarily, it should be checked whether there is any difference at all compared to the normal standard treatment by the doctors of the emergency department. For this, the different drug recommendations are compared.

For the qualitative evaluation, the second step is an analysis of the recommended drugs with regard to the use of inadequate preparations for older patients.

DETAILED DESCRIPTION:
Despite the changed age structure with a steady increase in life expectancy, doctors with geriatric expertise are lacking in many hospitals. In the "Rheinisch-Westfälische Technische Hochschule" (RWTH) Aachen University Hospital there is also the problem that the Department of Geriatrics is outsourced and therefore geriatric expertise is not always available in the emergency department. One way to solve this problem is to use telemedicine.

The aim of the present study is the implementation of a telemedical geriatric co-evaluation in the emergency department.

For the study it is planned to carry out a geriatric co-evaluation of geriatric emergency patients (age ≥ 70 years, "Identification of Seniors at Risk" [ISAR] -Score ≥ 2) with operative or conservative illnesses via a telemedical visit in the acute setting of the emergency department. There is a presentation of the patient by means of video transmission. The geriatrician then has the opportunity to question the patient independently or to carry out a physical assessment. Since there is no geriatrician at the Department of Geriatrics 24 hours a day, patients are included on weekdays between 8am and 5pm only.

Whenever possible, all patients in the emergency department at this time with an age ≥ 70 years and an ISAR score ≥ 2 will be enrolled at set times of the day. Due to the high number of patients in the emergency room, however, it may not be possible at times to include all patients. In order to ensure sufficient neutrality, in this constellation, the selection is made from the patients currently in the emergency room by means of randomization. Should there be age-related difficulties in communicating between patients and geriatrician during the telemedical visit, the present scientific assistant or doctor from the emergency department will assist to avoid an associated influence on the procedure.

The rationale behind the telemedicine visit is that this additional early geriatric co-assessment will result in improved geriatric follow-up beyond geriatric special care. In this pilot study, which aims at an analysis of the actual state with identification of potential problem areas, the focus is primarily on pharmacotherapeutic aspects.

The aim is to compare the diagnostic and treatment recommendations initiated in the emergency room by means of telemedical geriatric consultation with the standard treatment of the treating internist, neurologist or surgical assistant doctors of the central emergency department. The treatment plan defined in the telemedical visit is only a treatment recommendation. Prior to the implementation of the recommendations, a check is carried out by the responsible senior physician of the emergency department after completing the emergency geriatric visit. Thus, there are no risks dependent on the procedure for the patient.

Due to the high priority of the drug therapy in the emergency department, the primary endpoint is a comparison of the drug recommendations. Initially, a quantitative evaluation with determination of the number of different views per patient in the pharmacological differential therapy was performed. Secondary endpoints are to evaluate the use of medications that are considered inadequate for elderly patients. Since no special list of inadequate drugs has been validated specifically for the emergency room, the treatment recommendations are checked using a standard treatment list, the "Fit for the aged" (FORTA) classification system.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 70 years
* Written declaration of consent
* Indication for geriatric treatment according to "Identification of Seniors at risk" (ISAR) score screening with scores ≥ 2
* Persons who are capable and mentally able to follow the instructions of the study staff
* Legally incompetent persons with a consensual legal guardian or a person authorized by the patient to manage their affairs

Exclusion Criteria:

* Persons who are accommodated on an official or court order in an institution
* Persons who are in a dependency or employment relationship with the sponsor or examiner
* Simultaneous participation in another clinical trial
* Missing written consent

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Geriatric emergency patients aged ≥ 70, who showed an "Identification of Seniors at risk"-Score (ISAR-Score) ≥ 2.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Differences in pharmacological interventions | within 48 hours of admission to the emergency department
  The primary endpoint is an evaluation of the different pharmaceutical interventions between the standard emergency department treatment and the telemedicine geriatric treatment.
  Number of different views per patient in the pharmacological differential therapy with regard to:
  * drug replacement
  * withdrawal of a pre-existing drug
  * dose adjustment of a pre-existing drug are being analyzed.

SECONDARY OUTCOMES:
Quality of pharmacological interventions | within 48 hours of admission to the emergency department
  The secondary endpoint is an evaluation of the different pharmacological interventions with a focus on age-appropriate adequate medication. The treatment recommendations were checked with the FORTA classification system.
Avoidance of Polypharmacy as a quality feature for age-appropriate therapy | within 48 hours of admission to the emergency department
  Another secondary endpoint is an examination of the treatment recommendations regarding especially the reduction of total medication. Polypharmacy, as well as the use of inadequate drugs in geriatric patients, is a risk factor for complications.

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Brokmann, PD Dr., Study Director — Emergency Department, University Hospital RWTH Aachen, Aachen, Germany
Locations (1):
- Emergency department, University Hospital RWTH Aachen, Aachen, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Werner H. [Drug therapy in the aged: too much and too little, what to do? A new evaluation system: fit for the aged (FORTA)]. Dtsch Med Wochenschr. 2009 Jan;134(3):95-6; author reply 96. doi: 10.1055/s-0028-1105898. Epub 2009 Jan 13. No abstract available. German. PMID 19142841
- [Background] Yao JL, Fang J, Lou QQ, Anderson RM. A systematic review of the identification of seniors at risk (ISAR) tool for the prediction of adverse outcome in elderly patients seen in the emergency department. Int J Clin Exp Med. 2015 Apr 15;8(4):4778-86. eCollection 2015. PMID 26131052
- [Derived] Matz O, Villa L, Lecce C, Olaciregui Dague K, Haeger A, Bollheimer LC, Laurentius T, Rossaint R, Brokmann J. Implementation of a telemedicine geriatric co-evaluation in the emergency department: a prospective pilot study. Swiss Med Wkly. 2021 May 5;151:w20500. doi: 10.4414/smw.2021.20500. eCollection 2021 Apr 26. PMID 34000061